CLINICAL TRIAL: NCT00014872
Title: Genetic Epidemiology and Energy Metabolism in Black Girls
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently entered into CT.gov
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 968; R01HL066070 (NIH)
Record Dates: First submitted 2001-04-11; First posted 2001-04-12 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To investigate the role of genes and energy metabolism in the pathogenesis of obesity in adolescent Black girls.

DETAILED DESCRIPTION:
BACKGROUND:

The high prevalence of obesity in African-American (AA) women is of public health importance since AA women suffer higher mortality from cardiovascular and renal diseases than do white women. The reason for their marked susceptibility to obesity remains poorly understood though it is now known that AA women manifest lower resting energy expenditure than white women.

DESIGN NARRATIVE:

This is a multi-pronged metabolic and genetic epidemiologic study to examine two candidate genes (UCP3 and b3AR) implicated in energy metabolism. A total of 600 African American girls, aged 12-15 years, will be screened using buccal swabs as a non-invasive method of obtaining DNA, to determine their UCP3 genotypes as well as b3AR genotypes. An estimated 211 girls will be recruited, selected based on their UCP3 genotype, for measurements of resting energy expenditure and body composition (using dual energy X-ray absorptiometry [DEXA]) in a controlled setting of the Clinical Research Center at the Cincinnati Children's Hospital. Variation in resting energy expenditure will be examined across the genotypes of UCP3 with a large sample. The 2x3 design will allow the investigators to examine whether the effects associated with UCP3 variation are due to the UCP3 locus alone or due to the additive effect or interaction between UCP3 and b3AR. The study will help to elucidate the relationship between variation in two important candidate genes for energy metabolism, UCP3 and b3AR, and inter-individual variation in the levels of resting energy expenditure in this very high risk (for obesity) population.

ELIGIBILITY:
No eligibility criteria

Ages: 12 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: 12-15 years old black girl with Cardiovascular Diseases Obesity
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
UCP3 genotype correlation to obesity | six months

CONTACTS AND LOCATIONS:
Overall Officials: Sue Kimm, Principal Investigator — University of New Mexico